CLINICAL TRIAL: NCT00028587
Title: A Phase I and Pharmacologic Study of the Proteasome Inhibitor PS-341 in Combination With Paclitaxel and Carboplatin in Patients With Advanced Malignancies
Brief Title: PS-341 and Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02436; MC0012; CDR0000069108 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bortezomib; Paclitaxel; Taxes; Carboplatin

ARMS (2):
- Group I (paclitaxel, carboplatin, bortezomib) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and bortezomib IV over 3-5 seconds on days 2, 5, and 8.
  Interventions: Drug: bortezomib; Drug: paclitaxel; Drug: carboplatin; Other: laboratory biomarker analysis
- Group II (bortezomib, paclitaxel, carboplatin) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, and 8 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 2
  Interventions: Drug: bortezomib; Drug: paclitaxel; Drug: carboplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
Phase I trial to study the effectiveness of combining PS-341 and combination chemotherapy in treating patients who have advanced solid tumors. PS-341 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining PS-341 and chemotherapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of bortezomib and paclitaxel administered in combination with carboplatin in patients with advanced solid tumors.

II. Compare the tolerability and efficacy of the different sequences of this regimen in these patients.

III. Determine the clinical toxic effects and pharmacokinetics of this regimen in these patients.

IV. Determine, preliminarily, the therapeutic activity of this regimen in these patients.

V. Evaluate p53 accumulation as a marker of PS-341 activity, and the effect of paclitaxel/carboplatin on PS-341 induced accumulation of p53.

VI. Exam the effect of PS-341 on the levels of other proteasome targets, e.g. mdm2, p27, p21, cyclins B, D1,E; IκB and other ubiquitinated proteins in tumor tissue, when available.

OUTLINE: This is a dose-escalation study of bortezomib and paclitaxel. Patients are assigned to 1 of 2 treatment groups.

Group A: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and bortezomib IV over 3-5 seconds on days 2, 5, and 8.

Group B: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, and 8 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 2.

Treatment in both groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. After 6 courses of paclitaxel and carboplatin, patients with stable or responding disease may continue with bortezomib alone at the discretion of the investigator. Cohorts of 3-6 patients in each group receive escalating doses of bortezomib and paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 months.

PROJECTED ACCRUAL: A total of 24-96 patients will be accrued for this study within 25 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy for which no known standard therapy that is potentially curative or definitely capable of extending life expectancy exists
* No hematologic malignancies
* No symptomatic CNS metastases

  * Brain metastases allowed if previously treated (radiotherapy and/or surgery)and patient is stable for at least 8 weeks
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No New York Heart Association class III or IV heart disease
* HIV negative
* No peripheral neuropathy grade 2 or greater
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior immunotherapy
* No prior bone marrow transplantation
* No concurrent immunotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 30% of bone marrow
* No concurrent radiotherapy
* No concurrent investigational ancillary therapy
* No concurrent enrollment in another study involving a pharmacologic agent (e.g., drugs, biologics, immunotherapy, or gene therapy) for symptom control or therapeutic intents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2001-12; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
MTD of paclitaxel, bortezomib, and carboplatin defined as the highest safely-tolerated dose where =< 1 patient experience dose-limiting toxicity (DLT) with the next higher dose having at least 2 patients who experience DLT as assessed by CTC version 2.0 | 21 days
Number of toxicity incidents as assessed by CTC Version 2.0 | 21 days
  Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Number of responses | Up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses.
Change in p53 accumulation | From baseline to up to 3 months
Change in other proteasome levels | From baseline to up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States